CLINICAL TRIAL: NCT00068692
Title: Intergroup Randomized Phase III Study of Postoperative Irinotecan, 5-Fluorouracil and Leucovorin vs. Oxaliplatin, 5-Fluorouracil and Leucovorin vs. 5-Fluorouracil and Leucovorin for Patients With Stage II or III Rectal Cancer Receiving Either Preoperative Radiation and 5-Fluorouracil or Postoperative Radiation and 5-Fluorouracil
Brief Title: Comparison of Adjuvant Chemotherapy Regimens in Treating Stage II/III Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02959; NCI-2012-02959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E3201 (Other: ECOG-ACRIN Cancer Research Group); U10CA021115 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Rectal Mucinous Adenocarcinoma; Rectal Signet Ring Cell Adenocarcinoma; Recurrent Rectal Carcinoma; Stage IIA Rectal Cancer AJCC v7; Stage IIB Rectal Cancer AJCC v7; Stage IIC Rectal Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7; Stage IVA Rectal Cancer AJCC v7; Stage IVB Rectal Cancer AJCC v7
Keywords: rectal cancer; chemotherapy; irinotecan; oxaliplatin
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Fluorouracil; Leucovorin; Oxaliplatin; Platinum; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group I, Arm I (Experimental): Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Irinotecan
- Group I, Arm II (Experimental): Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 8 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin
- Group I, Arm III (Experimental): Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 1 hour on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 8 weeks for 3 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium
- Group II, Arm I (Experimental): Patients receive irinotecan, leucovorin calcium, and fluorouracil as in group 1, arm I for 4 courses. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Irinotecan
- Group II, Arm II (Experimental): Patients receive oxaliplatin, leucovorin calcium, and fluorouracil as in group 1, arm II for 4 courses. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Drug: Oxaliplatin
- Group II, Arm III (Experimental): Patients receive leucovorin calcium and fluorouracil as in group 1, arm III for 1 course. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiotherapy; Drug: Fluorouracil; Drug: Leucovorin Calcium

INTERVENTIONS:
Radiation: Radiotherapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; external radiation
Drug: Fluorouracil — Given IV
  Other Names: Efudex; 5-FU; 5-Fluorouracil; Adrucil
Drug: Leucovorin Calcium — Given IV
  Other Names: Leucovorin; Wellcovorin; citrovorun factor; folinic acid; LV; LCV; 5-formyl tetrahydrofolate
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacplat; Eloxatin; Eloxatine; Trans-l-diaminocyclohexane oxalatoplatinum; Cis-[oxalato (trans-I-1 ,2-diaminocyclohexane) platinum(lI)]; cis -[(1R,2R)-1,2-cyclohexanediamine- N,N'] [oxalate(2-)- 0,0'] platinum
  Arms: Group I, Arm II; Group II, Arm II
Drug: Irinotecan — Given IV
  Other Names: Camptosar; CPT-11; Camptothecin-11
  Arms: Group I, Arm I; Group II, Arm I

SUMMARY:
This randomized phase III trial is comparing the effectiveness of three adjuvant combination chemotherapy regimens in treating patients who are receiving radiation therapy and fluorouracil either before or after surgery for stage II or stage III rectal cancer. Drugs used in chemotherapy, such as irinotecan, fluorouracil, leucovorin, and oxaliplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which adjuvant combination chemotherapy regimen is more effective in treating patients who are receiving radiation therapy and fluorouracil either before or after surgery for rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival of patients treated with irinotecan, 5-FU and leucovorin versus those treated with oxaliplatin, leucovorin and 5-FU versus those treated with leucovorin and 5-FU for patients with stage II and III rectal cancer.

SECONDARY OBJECTIVES:

I. To determine sphincter preservation, tolerance of treatment and patterns of failure.

II. To describe patterns of failures

OTHER PRE-SPECIFIED OBJECTIVES:

I.To prospectively assess rectal function using the Patient Bowel Function/Uniscale questionnaire and the FACT Diarrhea Subscale in patients treated with an adjuvant program of pelvic radiation therapy and chemotherapy.

II. To correlate expression of key targets for 5-FU, leucovorin, oxaliplatin and irinotecan from tumor tissue biopsies with treatment efficacy III. To correlate tumor molecular prognostic markers with survival. IV. To determine physician preference in regard to the radiation-chemotherapy sequence in the Intergroup.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1), chemotherapy/radiotherapy sequence (preoperative vs postoperative), and risk group (high risk [T3, N+, M0 or T4, any N, M0] vs low risk [T1-2, N+, M0 or T3, N0, M0]). Patients are treated in 1 of 2 groups according to physician preference and then randomized to 1 of 3 treatment arms.

GROUP I (preoperative chemoradiotherapy and additional adjuvant chemotherapy): Preoperative chemoradiotherapy: Patients receive 1 of 3 treatment regimens, determined by the treating physician.

REGIMEN A (radiotherapy and fluorouracil): Patients undergo external beam radiotherapy once daily 5 days a week for 5 1/2 weeks (total of 28 fractions). Patients also receive concurrent fluorouracil intravenously (IV) continuously 7 days a week for 5 1/2 weeks.

REGIMEN B (radiotherapy, fluorouracil, and leucovorin calcium): Patients undergo external beam radiotherapy as in regimen A. Patients also receive concurrent fluorouracil IV and leucovorin calcium IV continuously for 4 days on weeks 1 and 5.

REGIMEN C (radiotherapy and capecitabine)*: Patients undergo external beam radiotherapy as in regimen A. Patients also receive concurrent oral capecitabine twice daily for 5 1/2 weeks.

NOTE: *Regimen C is allowed only for patients enrolled on protocol NSABP-R-04.

Surgery: Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection.

Additional adjuvant chemotherapy: Within 21-56 days after complete surgical resection, patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 8 courses.

ARM II: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 8 courses.

ARM III: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 1 hour on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 8 weeks for 3 courses.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

GROUP 2 (postoperative chemoradiotherapy and additional adjuvant chemotherapy): Within 21-56 days after complete surgical resection, patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive irinotecan, leucovorin calcium, and fluorouracil as in group 1, arm I for 4 courses.

ARM II: Patients receive oxaliplatin, leucovorin calcium, and fluorouracil as in group 1, arm II for 4 courses.

ARM III: Patients receive leucovorin calcium and fluorouracil as in group 1, arm III for 1 course.

Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemoradiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually for 5 years.

ELIGIBILITY:
1. Group I (Pre-operative) Registration

   Inclusion Criteria:
   * Patients must have histologically proven adenocarcinoma of the rectum with no distant metastases. Clinical staging is required (T3N0M0, T4N0M0, TanyN1-3M0).
   * Patients must not have evidence of tumor outside of the pelvis including liver metastases, peritoneal seeding, or metastatic inguinal lymphadenopathy.
   * The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 cm of anal verge by proctoscopic examination. In addition, patients who have had a portion of their tumors confirmed to be below the peritoneal reflection at the time of surgery are eligible regardless of the distance determined by endoscopy.
   * Transmural penetration of tumor through the muscularis propria must be demonstrated by CT scan, endo-rectal ultrasound or MRI.
   * Tumors must be defined prospectively by the surgeon as clinically resectable or not.

     * Clinically resectable tumors will be defined by the surgeon as not fixed and completely resectable with negative margins based on the routine examination of the non-anesthetized patient.
     * Before pre-op treatment, the surgeon should estimate and record the type of resection anticipated: APR, LAR or LAR/coloanal anastomosis.
   * The tumor may be clinically fixed or initially not completely resectable, clinical stage T4 N0-2 M0 based on the presence of at least one of the following criteria:

     * Clinically fixed tumors on rectal examination with tumor adherent to the pelvic sidewall or sacrum.
     * Hydronephrosis on CT scan or IVP or ureteric or bladder invasion as documented by cystoscopy and cytology or biopsy, or invasion into prostate.
     * Vaginal or uterine involvement.
   * Patients must not have a previous or concurrent malignancy, with the exception of:

     * Nonmelanoma skin cancer or in situ cervical cancer.
     * Treated non-pelvic cancer from which the patient has been continuously disease-free for >5 years.
   * Patients must have ECOG performance status 0-1.
   * Patients must be > 18 years of age.
   * All females of childbearing potential must have a blood or urine test within 2 weeks prior to registration to rule out pregnancy.
   * Sexually-active women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception

   Exclusion Criteria:
   * Patients have received prior chemotherapy or pelvic irradiation therapy.
   * Female patients must not be pregnant or breast-feeding.
   * Patients have an active inflammatory bowel disease or other serious medical illness which might limit the ability of the patient to receive protocol therapy.
2. Group II (Post-operative) Registration

   Inclusion Criteria:
   * Patients must have had histologically proven adenocarcinoma of the rectum with no distant metastases. Pathologic staging is required (T3N0M0, T4N0M0, TanyN1-3M0).
   * Patients must not have evidence of tumor outside of the pelvis including liver metastases, peritoneal seeding, or metastatic inguinal lymphadenopathy.
   * The distal border of the tumor must have been at or below the peritoneal reflection, defined as within 12 centimeters of anal verge by proctoscopic examination. In addition, patients who have had a portion of their tumors confirmed to be below the peritoneal reflection at the time of the surgery are eligible regardless of the distance determined by endoscopy.
   * Patients must not have received prior chemotherapy or pelvic irradiation therapy.
   * Patients must not have a previous or concurrent malignancy, with the exception of:

     * Non-melanoma skin cancer or in situ cervical cancer.
     * Treated non-pelvic cancer from which the patient has been continuously disease-free for >5 years.
   * Patients must have ECOG performance status 0-1.
   * Patients must be > 18 years of age.
   * All females of childbearing potential must have a blood or urine test within 2 weeks prior to registration to rule out pregnancy.
   * Sexually active women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.

   Exclusion Criteria:
   * Patients have an active inflammatory bowel disease or other serious medical illness which might limit the ability of the patient to receive protocol therapy.
   * Female patients are pregnant or breast-feeding.
3. Randomization (Groups I and II)

Inclusion Criteria:

* Patients must have a completely resected tumor and be within 21-56 days from the date of surgery.
* Patients who received combination chemotherapy/XRT prior to randomization (Group I) must have had a minimum radiation dose of 50.4 Gy.
* Patients must have ECOG performance status 0-1.
* Patients must have adequate renal function (creatinine < 1.5 x ULN) obtained < 4 weeks prior to randomization.
* Patients must have adequate hepatic function (bilirubin < 1.5 x ULN, SGOT (AST) < 3 x ULN) obtained < 4 weeks prior to randomization).
* Patients must have absolute neutrophil count > 1500/mm3 and platelet count > 100,000/mm3 < 4 weeks prior to randomization.

Exclusion Criteria:

• Patients have an active inflammatory bowel disease or other serious medical illness which might limit the ability of the patient to receive protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2003-10-15; Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Benson, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared upon approval

REFERENCES:
- [Derived] Kam AE, Zhao F, Meropol NJ, Giantonio BJ, Diasio RB, Flynn PJ, Catalano P, Hartner L, Rowland KM, Song W, Mulcahy MF, Sinicrope FA, Whitehead RP, Mayer RJ, Petrelli N, O'Dwyer PJ, Hamilton SR, Cella D, Benson AB. Intergroup randomized phase III study of adjuvant FOLFIRI, FOLFOX, or 5-FU/leucovorin for stage II/III rectal cancer: ECOG-ACRIN E3201. Oncologist. 2025 Dec 27;31(1):oyaf416. doi: 10.1093/oncolo/oyaf416. PMID 41397917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on October 15, 2003. Accrual was suspended on November 26, 2004 and subsequently closed on October 25, 2005 with total accrual of 225 patients to step 1 and 179 patients to step 2.
Groups:
- Group I, Arm S: Group I patients receive concurrent chemotherapy and radiation prior to surgery.
- Group II, Arm T: Patients who had surgery before registering to the study was in Group II. They were registered and randomized at the same time.
- Group II, Arm I: Patients receive irinotecan, leucovorin calcium, and fluorouracil as in group 1, arm I for 4 courses. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy
  Fluorouracil: Given IV
  Leucovorin Calcium: Given IV
  Irinotecan: Given IV
- Group II, Arm II: Patients receive oxaliplatin, leucovorin calcium, and fluorouracil as in group 1, arm II for 4 courses. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy
  Fluorouracil: Given IV
  Leucovorin Calcium: Given IV
  Oxaliplatin: Given IV
Period: Step 1: Registration
Arm/Group | Group I, Arm S | Group II, Arm T | Group I, Arm I | Group I, Arm II | Group I, Arm III | Group II, Arm I | Group II, Arm II | Group II, Arm III
Started (Randomization (arms I-III in both groups) was step 2.) | 128 | 97 (Group II patients were registered and randomized at the same time, and were reported in Step 2.) | 0 | 0 | 0 | 0 (Group II patients was registered and randomized at the same time, and reported in step 2) | 0 (Group II patients was registered and randomized at the same time, and reported in step 2) | 0 (Group II patients was registered and randomized at the same time, and reported in step 2)
Started Concurrent Chemo/Radiation | 125 | 0 (Group II patients receive protocol therapy in Step 2 after randomization) | 0 | 0 | 0 | 0 | 0 | 0
Reported AE Data | 123 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Of the 88 patients completed step 1 treatment, 5 of them decided not to randomize to step 2) | 88 | 96 (Case 32191 entered the study as Group II patient but was never randomized.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 40 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disese progression/relapse | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Alternative therapy | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Complicating disease | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not eligible | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not start protocol therapy | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Registered but not randomized | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2: Randomization
Arm/Group | Group I, Arm S | Group II, Arm T | Group I, Arm I | Group I, Arm II | Group I, Arm III | Group II, Arm I | Group II, Arm II | Group II, Arm III
Started (Randomization (arms I-III in both groups) was step 2.) | 0 (Patients on arm S completing step 1 treatment were randomized to step 2 (Arms I-III).) | 0 (Group II patients were registered and randomized at the same time, reported as arms I,II,III here.) | 28 (Of the 128 patients registered to step 1in group 1, 83 were randomized to step 2(arms I-III).) | 25 (Of the 128 patients registered to step 1in group 1, 83 were randomized to step 2(arms I-III).) | 30 (Of the 128 patients registered to step 1in group 1, 83 were randomized to step 2(arms I-III).) | 31 (Group 2 patients were registered and randomized at the same time.) | 33 (Group 2 patients were registered and randomized at the same time.) | 32 (Group 2 patients were registered and randomized at the same time.)
Treated | 0 | 0 | 27 | 25 | 29 | 31 | 33 | 32
Had Sphincter Preservation | 0 | 0 | 28 | 25 | 28 | 31 | 33 | 30
Reported AE Data | 0 | 0 | 27 | 22 | 28 | 31 | 33 | 32
Completed | 0 | 0 | 18 | 13 | 21 | 25 | 29 | 24
Not Completed | 0 | 0 | 10 | 12 | 9 | 6 | 4 | 8
Not completed — Disesae progression/replase | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 2 | 2 | 3 | 4 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 6 | 3 | 2 | 0 | 3
Not completed — alternative therapy | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — never start protocol therapy | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients in Step 2
Groups:
- Irinocetan (Arm I): The study was not designed to look at the treatment regimen separately in the two groups. I in Group I and Group II are combined. Patients in this group received irinocetan plus 5-FU and leucovorin,
- Oxaliplatin (Arm II): The study was not designed to look at the treatment regimen separately in the two groups. I in Group I and Group II are combined. Patients in this group received oxaliplatin plus 5-FU and leucovorin.
- Control (Arm III): The study was not designed to look at the treatment regimen separately in the two groups. I in Group I and Group II are combined. Patients in this group only received 5-FU and leucovorin.
- Total: Total of all reporting groups
Arm/Group | Irinocetan (Arm I) | Oxaliplatin (Arm II) | Control (Arm III) | Total
Number analyzed (Participants) | 59 | 58 | 62 | 179
Age, Continuous [Median (Full Range); unit: years] | 58 [33 to 82] | 56 [35 to 79] | 58 [36 to 79] | 57 [33 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 19 | 60
  Male | 40 | 36 | 43 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 6
  White | 56 | 57 | 58 | 171
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival Rate
Description: Overall survival (OS) was defined as time from randomization to death from any cause. 3-year OS rate was estimated using Kaplan-Meier method.
Time Frame: assessed every 3 months withihn 2 years of study entry, every 6 monhts between years 3-5 and then annually for 5 years, estimated at 3 years
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Groups:
- Irinocetan (Arm I): The study was not designed to look at the treatment regimen separately in the two groups. I in Group I and Group II are combined. Patients in this group received irinocetan plus 5-FU and leucovorin.
Arm/Group | Irinocetan (Arm I) | Oxaliplatin (Arm II) | Control (Arm III)
Number analyzed (Participants) | 59 | 58 | 62
proportion of patients | 0.965 [0.868 to 0.991] | 0.843 [0.721 to 0.915] | 0.870 [0.757 to 0.933]
Statistical Analysis 1: Comparison: Irinocetan (Arm I) vs Control (Arm III); Test type: Superiority; p = 0.35, Log Rank — One-sided p value was reported; stratified on ECOG performance status, clinical stage, timing of chemoradiotherapy, and regimen administration
Statistical Analysis 2: Comparison: Oxaliplatin (Arm II) vs Control (Arm III); Test type: Superiority; p = 0.69, Log Rank — one-sided p value was reported; stratified on ECOG performance status, clinical stage, timing of chemoradiaotherapy, regimen administration

2. Secondary Outcome: 3-year Disease Free Survival
Description: Disease free survival (DFS) was defined as time from randomization to recurrence, second invasive primary cancer and death from any cause, whichever occurred first. 3-year DFS rate was estimated using Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Groups:
- Oxaliplatin (Arm II): The study was not designed to look at the treatment regimen separately in the two groups. I in Group I and Group II are combined.Patients in this group received oxaliplatin plus 5-FU and leucovorin.
Arm/Group | Irinocetan (Arm I) | Oxaliplatin (Arm II) | Control (Arm III)
Number analyzed (Participants) | 59 | 58 | 62
proportion of patients | 0.670 [0.533 to 0.776] | 0.717 [0.580 to 0.816] | 0.704 [0.572 to 0.802]

3. Secondary Outcome: Proportion of Sphincter Preservation
Description: Proportion of sphincter preservation was defined as number of patients with sphincter preservation divided by total number of patients randomized to the arm
Time Frame: assessed at primary surgery time
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Irinocetan (Arm I) | Oxaliplatin (Arm II) | Control (Arm III)
Number analyzed (Participants) | 59 | 58 | 58
proportion of patients | 0.814 [0.691 to 0.903] | 0.724 [0.591 to 0.833] | 0.655 [0.519 to 0.775]

4. Secondary Outcome: Failure Pattern
Description: Type of failures (local/regional recurrence vs. distant recurrence vs. concurrent recurrence vs. second primary cancer vs. deaths) in the analysis population
Time Frame: assessed every 3 months withihn 2 years of study entry, every 6 monhts between years 3-5 and then annually for 5 years
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Irinocetan (Arm I) | Oxaliplatin (Arm II) | Control (Arm III)
Number analyzed (Participants) | 59 | 58 | 62
Participants
  Local/regional recurrence only | 3 | 5 | 5
  Distant recurrence only | 15 | 11 | 10
  Both local/regional and distant recurrence | 2 | 4 | 1
  Any recurrence | 20 | 20 | 16
  Second primary cancer | 3 | 5 | 2
  Death | 19 | 21 | 21

ADVERSE EVENTS:
Time Frame: Assessed at the end of every cycle (1 cycle=2 weeks for Arm I and Arm II in both groups, 1 cycle=8 weeks for Arm III in both groups) while on treatment and for 30 days after the end of treatment, assessed up to 10 years
Description: Group 1 patients received concurrent chemotherapy and radiation in step 1, and then received the adjuvant therapy in step 2 after randomization. Adverse events were reported for step 1 (arm S) and step 2 (arms I,II,III) separately. Group 2 patients were registered and randomized at the same time, and adverse events for adjuvant therapy were reported at step 2 (arms I, II, III).
Groups:
- Arm S: Preoperative chemo/radiation therapy received by Group I patients in step 1
- Group I, Arm I: Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive irinotecan IV over 90 minutes and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy Fluorouracil: Given IV Leucovorin Calcium: Given IV Irinotecan: Given IV
- Group I, Arm II: Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours followed immediately by fluorourcil IV bolus on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for 8 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy Fluorouracil: Given IV Leucovorin Calcium: Given IV Oxaliplatin: Given IV
- Group I, Arm III: Patients receive 1 of 3 preoperative chemo and radiotherapy treatment regimens, determined by the treating physician. Within 21-56 days after the completion of chemoradiotherapy, patients undergo surgical resection. Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 1 hour on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 8 weeks for 3 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy Fluorouracil: Given IV Leucovorin Calcium: Given IV
- Group II, Arm III: Patients receive leucovorin calcium and fluorouracil as in group 1, arm III for 1 course. Within 4 weeks after the completion of chemotherapy, all patients undergo concurrent pelvic chemoradiotherapy as described in group 1 preoperative chemo and radiotherapy Regimen A, B, or C, followed 4-6 weeks later by 4 additional courses of adjuvant chemotherapy for arms I and II and 2 additional courses of adjuvant chemotherapy for arm III. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Radiotherapy: Undergo external beam radiation therapy Fluorouracil: Given IV Leucovorin Calcium: Given IV
Arm/Group | Arm S | Group I, Arm I | Group I, Arm II | Group I, Arm III | Group II, Arm I | Group II, Arm II | Group II, Arm III
All-Cause Mortality (participants affected / at risk) | 1/123 | 8/27 | 12/22 | 11/28 | 11/31 | 9/33 | 10/32
Serious Adverse Events (participants affected / at risk) | 62/123 | 11/27 | 14/22 | 10/28 | 21/31 | 23/33 | 23/32
Other Adverse Events (participants affected / at risk) | 27/123 | 7/27 | 3/22 | 3/28 | 6/31 | 6/33 | 12/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm S (N=123) | Group I, Arm I (N=27) | Group I, Arm II (N=22) | Group I, Arm III (N=28) | Group II, Arm I (N=31) | Group II, Arm II (N=33) | Group II, Arm III (N=32)
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0
Leukocytes decreased (Investigations) | 2 | 4 | 4 | 2 | 3 | 5 | 3
Lymphopenia (Investigations) | 8 | 0 | 4 | 1 | 2 | 0 | 1
Neutrophils decreased (Investigations) | 6 | 6 | 9 | 2 | 6 | 9 | 1
Platelets decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hematologic-other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac-ischemia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 8 | 2 | 0 | 3 | 3 | 0 | 4
Fever w/o neutropenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Radiation dermatitis (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 6 | 1 | 0 | 3 | 2 | 1 | 4
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 0 | 4 | 2 | 1 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 32 | 3 | 2 | 6 | 12 | 10 | 16
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Incontinence, anal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leak, incl. anastomotic, rectum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 | 0 | 1
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 8 | 0 | 0 | 0 | 0 | 0 | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muco/stomatitis (symptom) rectum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 0 | 2 | 2 | 1 | 3
Obstruction, colon (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 3 | 0 | 3
GI-other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Surgical hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection w/ gr3-4 neut, abdomen NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection w/ gr3-4 neut, pelvis NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection Gr0-2 neut, abdomen (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection Gr0-2 neut, catheter (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, penis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection Gr0-2 neut, rectum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection Gr0-2 neut, wound (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infection w/ unk ANC rectum (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection w/ unk ANC blood (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic/Laboratory-other (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdomen, pain (Gastrointestinal disorders) | 5 | 0 | 1 | 1 | 4 | 1 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head/headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathic, pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral cavity, pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectum, pain (Gastrointestinal disorders) | 6 | 0 | 0 | 0 | 1 | 0 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethra, pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain-other (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incontinence urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm S (N=123) | Group I, Arm I (N=27) | Group I, Arm II (N=22) | Group I, Arm III (N=28) | Group II, Arm I (N=31) | Group II, Arm II (N=33) | Group II, Arm III (N=32)
Anemia (Blood and lymphatic system disorders) | 15 | 7 | 3 | 1 | 2 | 2 | 4
Leukocytes decreased (Investigations) | 7 | 4 | 2 | 1 | 0 | 2 | 6
Neutrophils decreased (Investigations) | 0 | 4 | 1 | 0 | 2 | 2 | 2
Platelets decreased (Investigations) | 0 | 1 | 2 | 0 | 1 | 2 | 2
Fatigue (General disorders) | 13 | 3 | 3 | 1 | 3 | 4 | 8
Weight loss (Investigations) | 8 | 0 | 0 | 0 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 0 | 1 | 2
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 10 | 4 | 1 | 1 | 3 | 3 | 5
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 7 | 1 | 0 | 0 | 2 | 1 | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 10 | 4 | 3 | 1 | 1 | 3 | 6
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 2
Abdomen, pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-06-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT00068692/Prot_SAP_000.pdf